CLINICAL TRIAL: NCT00648817
Title: A Phase IV, Randomized, Double-Blind, Placebo-Controlled, Two-Phase Crossover Study of the Metabolic Impact of Tenofovir Disoproxil Fumarate on HIV-1 Seronegative Healthy Adult Males
Brief Title: Metabolic Impact Assessment of Tenofovir Disoproxil Fumarate on Non-HIV-1 Infected Healthy Adult Male Volunteers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-104-0318; EUDRACT Number: 2004-005083-25
Record Dates: First submitted 2008-03-27; First posted 2008-04-01 (Estimated); Last update posted 2008-04-01 (Estimated); Status verified 2008-03

CONDITIONS: HIV Infections
Keywords: HIV-1; tenofovir DF
MeSH Terms: conditions — HIV Infections | interventions — Tenofovir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Placebo Comparator): * Tenofovir DF 300 mg QD (equivalent to 245 mg of tenofovir disoproxil) for the first 14 days of the study.
  * Tenofovir DF placebo tablet QD for the last 14 days of the study.
  Interventions: Drug: Tenofovir Disoproxil Fumarate; Drug: Tenofovir DF placebo
- Group 2 (Active Comparator): * Tenofovir DF placebo tablet QD for the first 14 days of the study.
  * Tenofovir DF 300 mg QD (equivalent to 245 mg of tenofovir disoproxil) for the last 14 days of the study.
  Interventions: Drug: Tenofovir Disoproxil Fumarate; Drug: Tenofovir DF placebo

INTERVENTIONS:
Drug: Tenofovir Disoproxil Fumarate — Tenofovir DF 300 mg QD (equivalent to 245 mg of tenofovir disoproxil)
Drug: Tenofovir DF placebo — Tenofovir DF placebo tablet QD

SUMMARY:
Metabolic changes commonly occur in HIV therapy. The purpose of this study is to assess the impact on insulin sensitivity from the administration of tenofovir disoproxil fumarate 300 mg compared with placebo in non-HIV-1 infected healthy adult males. Additionally, endothelial function, adipocytokines and lipids will be monitored.

DETAILED DESCRIPTION:
Double-blind, randomized, placebo-controlled study using a two-sequence two-period crossover structure. Sixteen HIV-1-negative males will be randomized 1:1 to one of two treatment arms.

Group 1:

* Tenofovir DF 300 mg QD (equivalent to 245 mg of tenofovir disoproxil) for the first 14 days of the study.
* Tenofovir DF placebo tablet QD for the last 14 days of the study.

Group 2:

* Tenofovir DF placebo tablet QD for the first 14 days of the study.
* Tenofovir DF 300 mg QD (equivalent to 245 mg of tenofovir disoproxil) for the last 14 days of the study.

Physical examinations and laboratory analyses are conducted at screening, baseline, Day 14, and Day 28. A euglycaemic clamp protocol and an ECG are performed at the baseline, Day 14 and Day 28 visits.

The primary efficacy endpoint of this study is insulin-mediated glucose disposal during a hyperinsulinaemic euglycaemic clamp study. Endothelial function will be monitored by Selectin P/E and PAI-1 levels; adipocytokine levels will be monitored by measuring adiponectin and leptin levels; and lipid subfractions, including cholesterol (large and small subfractions of HDL and LDL) triglycerides and non-esterified fatty acids will be measured. Safety will be evaluated by adverse event and clinical laboratory test reporting.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have documented negative HIV serology by ELISA and P24 antigen. This will be done at the screening visit.
* Subjects must be clinically well males aged between 18 to 55 years.
* Adequate renal function:
* Calculated creatinine clearance (CrCl) >= 100 mL/min according to the Cockcroft Gault formula: Male: [(140 - age in years) x (actual body wt in kg)]/[72 x (serum creatinine in mg/dL)]= CrCl (mL/min)
* Fasting blood glucose, total cholesterol and triglycerides within normal limits
* Hepatic transaminases (AST and ALT) <= 3 x upper limit of normal (ULN)
* Total bilirubin <= 1.5 mg/dL
* Adequate hematologic function (absolute neutrophil count >= 1,000/mm3; platelets >= 50,000/mm3; hemoglobin >= 8.0 g/dL)
* Serum amylase <= 1.5 x ULN (subjects with serum amylase > 1.5 x ULN will remain eligible if pancreatic lipase is <= 1.5 x ULN)
* Serum phosphorus >= 2.2 mg/dL
* Sexually active males must use condoms
* Life expectancy >= 1 year
* The ability to understand and sign a written informed consent form, which must be obtained prior to initiation of study procedures

Exclusion Criteria:

* Subjects with a waist hip ratio > 0.97 or BMI > 28 kg/m2 will be excluded
* Acute or chronic hepatitis B infection (determined by positive hepatitis B surface antigen result at the screening visit)
* Acute or chronic hepatitis C infection (determined by positive hepatitis C antibody result at the screening visit)
* Other metabolic syndrome or disease process likely to cause marked disturbance in glucose and lipid homeostasis
* Receiving on-going therapy with any of the following:
* Metabolically active medications
* Any lipid-lowering medication

  * Hormonal agents (oestrogens or androgens)
  * Glucocorticoids
  * Beta-blockers
  * Thiazide diuretics
  * Thyroid preparations
  * Psychotropic agents
  * Anabolic steroids
  * Megoestrol acetate
  * Nephrotoxic agents

    * aminoglycoside antibiotics
    * IV amphotericin B
    * cidofovir
    * cisplatin
    * foscarnet
    * IV pentamidine
    * other agents with significant nephrotoxic potential
  * Vancomycin
  * Oral or IV ganciclovir
  * Agents that inhibit or compete for elimination via active renal tubular secretion

    ** Probenecid
  * Systemic chemotherapeutic agents (i.e., cancer treatment medications)
  * Systemic corticosteroids
  * Interleukin 2 (IL 2) and other immunomodulating agents
  * Investigational agents

Administration of any of the above medications must be discontinued at least 30 days prior to the baseline visit and for the duration of the study period.

* Evidence of a gastrointestinal malabsorption syndrome or chronic nausea or vomiting which may confer an inability to receive an orally administered medication.
* Current alcohol or substance abuse judged by the investigator to potentially interfere with subject compliance.
* Malignancy or basal cell carcinoma.
* Active, serious infections requiring parenteral antibiotic therapy within 15 days prior to screening.
* Prior history of significant renal or bone disease.
* Subjects should avoid giving blood for the duration of this study.
* Any other clinical condition or prior therapy that, in the opinion of the investigator, would make the subject unsuitable for the study or unable to comply with the dosing requirements.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2006-07; Primary Completion 2007-11 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
To assess the impact on insulin sensitivity (determined by peripheral glucose uptake suing a euglycaemic clamp) of the administration of tenofovir DF compared with placebo for two weeks in HIV-1 seronegative healthy male volunteers.

SECONDARY OUTCOMES:
To assess endothelial function by monitoring changes in Selectin P/E and PAI-1 assays.
To monitor adipocytokines by assessing adiponectin and leptin levels.
To monitor lipids by assessing large and small lipoprotein sub-fractions of HDL and LDL cholesterol, triglycerides, and non esterified fatty acid concentrations.

CONTACTS AND LOCATIONS:
Overall Officials: Graeme Moyle, MD, MB, BS, DipGUM, Principal Investigator — Chelsea and Westminster Hospital, London, UK
Locations (1):
- Chelsea and Westminster Hospital, London, United Kingdom